CLINICAL TRIAL: NCT02128906
Title: A Randomized, Phase II Study of Definitive Radiotherapy With Concurrent Cisplatin vs. Docetaxel-cetuximab in Locally Advanced Head and Neck Squamous Cell Carcinoma: an ERCC1 Biomarker Enrichment and Interaction Design
Brief Title: Radiotherapy With Cisplatin vs. Docetaxel-cetuximab in HNSCC: ERCC1 Biomarker Enrichment and Interaction Design
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christopher Wilke (Other)
Responsible Party: Sponsor-Investigator, Christopher Wilke, Radiation Oncologist, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 13-056
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Squamous Cell Carcinoma
Keywords: ERCC1; oropharynx; larynx; hypopharynx; p16; radiotherapy; docetaxel; cetuximab; cisplatin; EGFR; head and neck
MeSH Terms: conditions — Carcinoma, Squamous Cell; Laryngeal Diseases | interventions — Cisplatin; Docetaxel; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cisplatin-IMRT (Active Comparator): Cisplatin 40 mg/m2 weekly x 7; IMRT: once daily, M-F, 7 weeks (70 Gy)
  Interventions: Drug: Cisplatin; Radiation: IMRT
- Docetaxel-Cetuximab-IMRT (Active Comparator): Docetaxel 15 mg/m2 weekly x 7; Cetuximab 400 mg/m2 load, one week prior to IMRT; Cetuximab 250 mg/m2 weekly x 7; IMRT: once daily, M-F, 7 weeks (70 Gy)
  Interventions: Radiation: IMRT; Drug: Docetaxel; Drug: Cetuximab

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 40 mg/m2 weekly x 7
  Other Names: Platinol
  Arms: Cisplatin-IMRT
Radiation: IMRT — IMRT: once daily, M-F, 7 weeks (70 Gy)
Drug: Docetaxel — Docetaxel 15 mg/m2 weekly x 7
  Other Names: Taxotere
  Arms: Docetaxel-Cetuximab-IMRT
Drug: Cetuximab — Cetuximab 400 mg/m2 load, one week prior to IMRT Cetuximab 250 mg/m2 weekly x 7
  Other Names: Erbitux
  Arms: Docetaxel-Cetuximab-IMRT

SUMMARY:
The goal of this clinical research study is to learn which chemotherapy combination may be more effective in treating locally advanced head and neck squamous cell carcinoma (HNSCC). The side effects of these combinations will also be studied.

This study treatment consists of intensity-modulated radiation therapy (IMRT) and concurrent chemotherapy. For study chemotherapy, patients will be randomized between cisplatin or the combination of docetaxel and cetuximab. Subjects will be stratified depending on HPV status and the presence of ERCC-1 [4F9] in the tumor prior to randomization. The study will evaluate cisplatin vs. docetaxel-cetuximab in the overall population, and test which radiation and chemotherapy combination works best in relationship to how much ERCC-1 [4F9] is expressed in a tumor.

DETAILED DESCRIPTION:
If randomized to the cisplatin arm, patients receive cisplatin, 40 mg/m2, administered intravenously (IV) once a week (+/- 2 days) for 7 weeks. Per investigator discretion, if radiation continues beyond 7 weeks due to technical factors (not toxicity delays), an 8th dose of concurrent cisplatin may be added.

Cisplatin can be given either before or after the radiation therapy fraction that is given on the same day. If a dose of cisplatin is omitted when radiotherapy is ongoing, it will not be made up or added to the end of treatment. The omitted dose and the reason for the omission should be recorded in the site's source documentation. If radiotherapy is held, cisplatin should be held during the treatment break and resumed when radiation restarts.

Patients randomized to Cetuximab arm receive cetuximab, 250 mg/m2, IV over 60 minutes on a weekly schedule (+/- 2 days). . Cetuximab may be administered either before or after the radiation fraction that is given on the same day. Docetaxel will be administered at least 30 minutes following cetuximab. It is not permitted to make up missed doses of cetuximab or docetaxel. If a radiation therapy treatment break occurs, cetuximab should be held. When radiation restarts, cetuximab should resume.

Cetuximab will be given once a week (+/- 2 days) for a total of 7 doses concurrent with radiation therapy and docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed squamous cell carcinoma, undifferentiated carcinoma, or poorly differentiated carcinoma of the oropharynx, larynx, or hypopharynx with no evidence of distant metastasis. Biopsy sampling of primary tumor with pathology report documenting diagnostic tissue type is required.
* Patients must have stage III, IVa or IVb disease as determined by imaging studies and complete head and neck exam. Staging evaluation should be in accordance with the American Joint Committee on Cancer Staging Manual, 7th edition.
* Patients with oropharyngeal squamous cell carcinoma may have p16(+) or p16(-) disease; in these patients, p16 status must be known prior to randomization. Assessment of p16 status may occur locally or centrally. Note: The definition of p16(+) disease is diffuse nuclear and cytoplasmic staining in ≥ 70% of tumor cells.
* Patients must be untreated with curative-intent surgery for current diagnosis of Stage III, IVa, or IVb disease. Diagnostic biopsy of primary tumor and/or nodal sites is permitted.
* Diagnostic simple tonsillectomy is permitted, provided patient has RECIST-measurable residual tumor and/or nodal disease.
* Patients with a second HNSCC primary tumor are eligible for this study, provided more than 2 years have elapsed since the first diagnosis of HNSCC, the original tumor was managed with surgery only (no adjuvant chemotherapy/radiotherapy), and has not recurred.
* Patients with simultaneous primaries or bilateral tumors are excluded, with the exception of patients with bilateral tonsil cancers or patients with T1-2, N0, M0 resected differentiated thyroid carcinoma, who are eligible.
* No prior systemic treatment (chemotherapy or biologic/molecular targeted therapy) or radiation treatment for head and neck cancer.
* Patients may have received chemotherapy or radiation for a previous, curatively treated non-HNSCC malignancy, provided at least 2 years have elapsed.
* Patients must be untreated with radiation above the clavicles.
* Patients with a history of curatively-treated non-HNSCC malignancy must be disease-free for at least 2 years except for carcinoma-in-situ of cervix, non-melanomatous skin cancer, or T1-2, N0, M0 resected differentiated thyroid carcinoma.
* Diagnostic primary tumor tissue must be available for ERCC1 staining
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 (See Appendix 8)
* Age ≥ 18
* Patients must have measurable disease according to RECIST 1.1
* Patients must have the following laboratory values measured within 14 days of registration:
* Absolute neutrophil count (ANC) > 1500/mm3
* Hemoglobin (Hb) > 8.0 g/dL
* Platelet count (PLT) > 100,000/mm3
* Creatinine clearance ≥ 45 ml/min determined by 24-hour collection or estimated by the Cockraft-Gault formula:

Calculated Creatinine Clearance = [(140-age) X (actual body weight in kg) X (0.85 if female)]/(72 X serum creatinine)

* Serum bilirubin < 2 mg/dL
* AST (aspartate aminotransferase) and ALT (alanine aminotransferase) < 3 times upper limit of normal (ULN)
* The following assessments are required within 14 days prior to registration: Na, K, Cl, glucose, Ca, Mg, and albumin. The following metabolic values will exclude patients from study enrollment:
* Serum calcium (ionized or adjusted for albumin) < 7 mg/dl (1.75 mmol/L) or > 12.5 mg/dl (> 3.1 mmol/L) despite intervention to normalize levels
* Magnesium < 0.9 mg/dl (< 0.4 mmol/L) or > 3 mg/dl (> 1.23 mmol/L) despite intervention to normalize levels
* Potassium < 3.5 mmol/L or > 6 mmol/L despite intervention to normalize levels
* Sodium < 130 mmol/L or > 155 mmol/L despite intervention to normalize levels Note: Patients with an initial magnesium < 0.5 mmol/L (1.2 mg/dl) may receive corrective magnesium supplementation but should continue to receive either prophylactic weekly infusion of magnesium and/or oral magnesium supplementation (eg, magnesium oxide) at the investigator's discretion.
* No prior severe infusion reaction to a monoclonal antibody
* Written informed consent must be obtained from all patients prior to beginning therapy. Patients should have the ability to understand and the willingness to sign a written informed consent document.
* Informed consent must be obtained from all patients prior to beginning therapy, including consent for mandatory tissue submission for ERCC1 staining (and p16 staining if not locally conducted). Patients should have the ability to understand and the willingness to sign a written informed consent document.
* No unstable angina or myocardial infarction within the prior 6 months; no symptomatic congestive heart failure; no serious cardiac arrhythmia requiring medication; no cerebrovascular ischemia or stroke within the past 6 months.
* No uncontrolled intercurrent illness including active infection, uncontrolled diabetes, uncontrolled hypertension, or uncontrolled psychiatric illness which in the investigator's opinion would limit compliance with study requirements or compromise patient safety.
* Women must not be pregnant or breast feeding because chemotherapy and/or cetuximab may be harmful to the fetus or the nursing infant. Pregnant women are excluded from this study because chemotherapy and/or cetuximab have the potential for teratogenic or abortifacient effects.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while in this study, she should inform her treating physician immediately. All females of childbearing potential must have a blood test or urine study within 14 days of registration to rule out pregnancy.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible drug interactions with study drugs. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated. Note: HIV testing is not required for entry into this protocol.
* Patients may not be receiving any other anti-neoplastic investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-12-23 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Time To Progression (TTP) | Up to 5 years
  Time To Progression is the duration of time from date of study entry until the first appearance of new metastatic lesions or objective tumor progression in patients with increased tumoral ERCC1 expression. Progression is defined per RECIST v1.1 as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).

SECONDARY OUTCOMES:
Time to progression (TTP) | Up to 5 years
  Time To Progression is the duration of time from date of study entry until the appearance of new metastatic lesions or objective tumor progression in patients with decreased tumoral ERCC1 expression. Progression is defined per RECIST v1.1 as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Local Control Rate (LRC) | Up to 5 years
  Proportions of patients with a tumor volume equal to or less than the tumor volume at start of radiotherapy.
Rate of distant metastases | Up to 5 years
  Proportion of patients with new metastatic lesions or objective tumor progression in patients with increased tumoral ERCC1 expression. Progression is defined per RECIST v1.1 as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Validation candidate cutpoint | Up to 5 years
  Validation candidate cutpoint for decreased/normal vs. increased ERCC1 [4F9] expression in patients treated with cisplatin-IMRT. ERCC1 [4F9] expression is measured.
Response per RECIST 1.1 | Up to 5 years
  Proportion of patients that experience response to treatment per RECIST v1.1 Per RECIST v1.1: Complete Response(CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target)must have reduction in short axis to <10mm. Partial Response(PR): Atleasta30%decreaseinthesumof diameters of target lesions, taking as reference the baseline sum diameters.
2-year (Time to Progression) TTP | At 2 years
  Proportion of patients with new metastatic lesions or objective tumor progression in patients with increased tumoral ERCC1 expression. Progression is defined per RECIST v1.1 as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
FACT-H&N FACT - Head & Neck | Up to 2 years
  The FACT-H&N (version 4) consists of a cancer-specific questionnaire, FACT-G, in addition to 12 H&N cancer-specific items (the HN subscale). FACT-G is a 27-item measure that assesses general cancer quality of life. The FACT-G contains 4 subscales: physical, social/family, emotional, and functional well-being. Individuals are asked to indicate how true 27 statements are for them, using the past 7 days as the timeframe. Responses range from not at all (0), to very much (4) on a 5-point scale. Higher scores indicate better quality of life.
Functional Assessment of Cancer Therapy (FACT-Cog) | Up to 2 years
  The FACT-Cog consists of 37 questions exploring four different subscales of the cognitive function: perceived cognitive impairments (CogPCI: 20 items); perceived cognitive abilities (CogPCA: 9 items); comments from others (CogOth: 4 items); and the impact of perceived cognitive impairments on quality of life (CogQOL: 4 items). The patient must answer the questions by referring to the last seven days, expressing how many times a given situation has occurred during this period.The total FACT-Cog score is the sum of the four subscales and ranges from 0-148. The higher the total score, the better the cognitive function, and the lower the impact on patients' quality of life.
Patient Health Questionnaire (PHQ-9) | Up to 2 years
  The PHQ-9 is a 9-question, self-administered instrument used to screen for the presence and severity of depression. Patients score how frequently they have been bothered by symptoms over the past 2 weeks. Scores range from 0-27 with 0 being least depressed and 27 most depressed. Scores are also monitored for change in values from visit to visit. Any value above 5 is an indication of the necessity of treatment intervention.
General Anxiety Disorder-7 (GAD-7) | Up to 2 years
  GAD-7 is a self-administered questionnaire of seven items which measures the frequency of GAD symptoms. Patients are monitored for change in values from visit to visit.Scores range from 0-21; severity of anxiety increases in each escalation of 5 points. Higher scores indicate increased severity of depression.
Modified Edmonton Symptom Assessment System (MESAS) | Up to 2 years
  MESAS asks cancer patients or caregivers to score 9 common cancer symptoms (along with a 10th symptom of "other") on a scale of 0-10. The scores are transferred to a ESAS Graph, thereby allowing the practitioner to identify severity of each symptom at time of assessment. Each symptom is rated from 0-10 on a numerical scale with 0 indicating an absence of the symptom and 10 indicating the worst possible severity of the symptom.
Impact of Events Scale - Intrusion (IES-I) | Up to 2 years
  A self-administered, 7-item test used to evaluate the level of distress caused in patients by a traumatic event. The patient is asked to consider their experience with cancer during the past week and then rate how much they were bothered by the experience, from 0 (not at all) to 4 (extremely). This yields a score between 0 and 28. Higher scores indicate a greater intrusion or impact of distress in the patient's life due to cancer.
Disease Related Blame Scale (DBS) | Up to 2 years
  A self-administered 2-item quiz used to evaluate the level of blame patients are experiencing regarding their cancer. Asked to consider the extent to which they contributed to contracting cancer on a scale of 1 (not at all) to 5 (completely), patients answer the questions to generate a number between 2 and 10. The lower the number, the less self-incrimination the patient is enduring.
Perceived Threat Scale (PTS) | Up to 2 years
  PTS is used to measure the patient's belief regarding the level of threat cancer poses to his/her life. Three questions are asked and the patient answers on a scale of 1 (not at all) to 5 (extremely). A final score between 3 and 15 is generated; the higher the number, the more threatened the subject is by the cancer diagnosis.
The Brief Pain Inventory | Up to 2 years
  The Brief Pain Inventory - Short Form is a 9 item self-administered questionnaire to measure the severity of a person' pain in musculoskeletal conditions and its impact on the patient's daily function. Patients are to consider their pain over the past 24 hours and rate it on a 0 (no pain) to 10 (most severe pain) scale for each of the following points: its most severe, its least sever, its average and its appearance right now. Patients are also to provide a score between 0 (no relief) and 10 (complete relief) regarding the effectiveness of treatments or medicines in the past 24 hours. Finally, patients rate the amount of interference pain has in 7 basic life functions on a scale of 0-10 with 0 being "no effect" and 10 being "complete interference".

CONTACTS AND LOCATIONS:
Overall Officials: Christopher T Wilke, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center - Radiation Oncology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No